CLINICAL TRIAL: NCT07201311
Title: Reduction of Digestive Absorption of Toxic Substances by Combined Digestive Decontamination in Intensive Care - Randomized Single-center Study
Brief Title: Combined Gastrointestinal Decontamination in Acute Severe Poisoning
Acronym: DIMREATOX
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP231308; 2024-518739-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-09; First posted 2025-10-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Severe Poisoning With Cardiotropic or Psychotropic Drug; Admission to Intensive Care
Keywords: Poisoning; Cardiotropic drugs; Psychotropic drugs; Activated charcoal; Polyethylene glycol
MeSH Terms: conditions — Poisoning; Anthrax | interventions — Polyethylene Glycols

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled single-center clinical trial using open-label administration of the study drugs The intervention group will receive activated charcoal at the dose of 25-100g and serial activated charcoal 50g 6 times/day if sustained-release forms or drugs with enterohepatic circulation were ingested. Polyethylene glycol will be administered after activated charcoal at the maximum dose of 1L of polyethylene glycol/15kg of ideal body weight. Treatment with polyethylene glycol will be stopped if clear rectal effluent is observed before 24 hours and/or the maximum dose is reached.
  The standard treatment group will be treated according to the French guidelines with activated charcoal 25-100g and serial activated charcoal 50g 6 times/day if sustained-release forms or drugs with enterohepatic circulation were ingested.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined gastrointestinal decontamination (Experimental): Patients receive activated charcoal and polyethylene glycol
  Interventions: Drug: Combination of activated charcoal with polyethylene glycol for digestive decontamination
- Control - standard treatment group (Active Comparator): Patients receive activated charcoal according to French guidelines
  Interventions: Drug: Standard Treatment (Guideline-Based)

INTERVENTIONS:
Drug: Combination of activated charcoal with polyethylene glycol for digestive decontamination — A dose of 25-100g of activated charcoal via the nasogastric tube will be administered, followed by polyethylene glycol1L/15-20 kg ideal body weight at a flow rate of 1L/hour.
  polyethylene glycol will be continued until clear stools are obtained, a maximum of 24h of treatment of until the maximum dose of 1L per 15 kg of ideal body weight are administered.
  Serial activated charcoal 50g 6 times/day will be administered if prolonged-release forms or drugs with enterohepatic circulation were ingested.
  Arms: Combined gastrointestinal decontamination
Drug: Standard Treatment (Guideline-Based) — Patients receive activated charcoal according to French guidelines - activated charcoal 25-100g and serial activated charcoal 50g 6 times/day if sustained-release forms or drugs with enterohepatic circulation as routine treatment.
  Arms: Control - standard treatment group

SUMMARY:
Gastrointestinal absorption of high dose medication (toxicant) ingested under solid form for suicidal purposes, is prolonged in patients who need intensive care admission and mechanical ventilation. This is due to the large ingested amounts, slowed blood circulation in the digestive system due to low blood pressure, and the formation of conglomerates of pills (pharmacobezoars).

We make the hypothesis that combined decontamination of the digestive system with activated charcoal plus polyethylene glycol may reduce absorption of the ingested toxicant compared with standard care.

Two hundred patients requiring admission to intensive care and mechanical ventilation due to the effect of the ingested toxicant, will be included in a 1:1 randomized fashion over 24 months in the intervention group receiving combined decontamination and standard care group receiving activated charcoal according to guidelines.

The main objective is to show a decrease in the concentration of the toxicant after 24h of randomization.

DETAILED DESCRIPTION:
Rationale - digestive absorption of toxic substances ingested in solid form is prolonged in severely intoxicated patients admitted to intensive care and requiring intubation and mechanical ventilation. This prolonged absorption is favoured by the large quantity of tablets/pills ingested, the formation of pharmacobezoars, delayed formulations, co-ingestion of transit slowing agents (such as substances with an anticholinergic effect) and mesenteric hypoperfusion in the event of hypotension slowing absorption.

Digestive decontamination with activated charcoal combined with intestinal purging with polyethylene glycol (PEG) appears to be effective in pharmacokinetic studies, but its benefits have never been studied in intoxicated patients, particularly after admission to intensive care. Digestive decontamination using activated charcoal and polyethylene glycol could reduce toxic concentrations at 24 hours compared with the standard treatment group.

Main objective: To show the greatest reduction in the plasma concentration of the toxicant(s) (ingested parent molecules) at H24 of randomisation in the intervention group receiving activated charcoal + intestinal purge compared with the control group.

primary endpoint: Percentage change in the plasma concentration of the toxic substance(s) (ingested parent molecules) at 24 hours compared with its/their value(s) at randomisation.

Secondary objectives:

* To show the greater reduction in the plasma concentration of the toxic substance(s) (ingested parent molecules) at H48, H72 and H96 of randomisation in the intervention group compared with the control group;
* To demonstrate a reduction in the number of days of mechanical ventilation and the length of time spent in intensive care in the intervention group compared with the control group;
* To demonstrate the good tolerance of treatment by digestive decontamination in the intervention group.

Secondary endpoints:

* Percentage change in plasma concentration of toxicant(s) (ingested parent molecules) at H48, H72 and H96 compared with the value at randomisation
* Area under the concentration curve up to the 96th hour expressed as a percentage of the concentration at randomisation
* Number of days alive without mechanical ventilation for 28 days post-randomisation
* Number of days alive without resuscitation for 28 days post-randomisation
* Number of episodes of vomiting
* Number of ventilator-associated pneumonias
* Number of episodes of upper abdominal pain and diarrhoea;
* Presence of hypersensitivity reactions such as anaphylactic shock, angioedema, urticaria, rash and pruritus.

ELIGIBILITY:
Inclusion Criteria:

Patient aged ≥18, intoxicated and hospitalised in intensive care AND

* Main drug toxicant of functional type (any psychotropic or cardiotropic), adsorbable by activated charcoal And
* Main toxicant identified by the history taken by a healthcare professional on the ward or during care prior to the ward And
* Main toxicant identified within 3 hours of admission if the patient is already intubated on admission, or within 3 hours of intubation if the patient is intubated on the ward AND
* Patient intubated for effects attributed to the toxic agent (neuro-respiratory or haemodynamic failure) AND
* Patient with nasogastric tube or planned nasogastric tube and no contraindications AND
* Main toxicant whose assay can be performed by the toxicology laboratory at Lariboisière Hospital AND Inclusion according to the emergency clause
* Written informed consent from a parent/relative/trusted person. In the absence of a parent/relative/trusted person, the patient may be included under the emergency procedure and consent will be obtained as soon as possible.

Exclusion Criteria:

* No social security affiliation
* Non-intubated patient
* Contraindication to the administration of one of the study products (e.g. suspected digestive perforation, intestinal obstruction, inflammatory bowel disease, etc.)
* Inability to insert a nasogastric tube
* Repeated vomiting prior to inclusion, making digestive decontamination impossible
* Digestive haemorrhage in progress or during the previous month
* Ingestion of metals (e.g. iron, caesium, thallium, lead, copper, cadmium)
* Isolated or predominant alcohol poisoning (e.g. ethyl alcohol, ethylene glycol, methanol)
* Intoxication by gas (e.g. carbon monoxide or fire fumes)
* Intoxication by a caustic product (acids or bases)
* Main toxicant ingested under liquid form
* Intoxication by a toxic lesion
* Intoxication by a non-medicated product (e.g. party drugs)
* Intubation for causes not attributed to the ingested toxic substance (e.g. massive inhalation pneumonia)
* In-body carrier of drug pellets
* Pregnant or breast-feeding patients
* Patients being treated for dementia
* Patient under guardianship or curatorship
* Patients under legal protection
* Patients deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Percentage change in the plasma concentration of the toxic substance | 24 hours post-randomization
  The primary endpoint is the percentage change in the plasma concentration of the toxic substance at 24 hours compared with the value at randomization.
  The percentage variation is calculated as 100 x (Concentration at 24 hours post-randomization-Concentration at randomization)/ Concentration at randomization

SECONDARY OUTCOMES:
Percentage change in plasma concentration of toxicant | 48, 72 and 96 hours post-randomization
  The percentage variation is calculated as:
  At 48 hours : 100 x (Concentration at 48 hours post-randomization-Concentration at randomization)/ Concentration at randomization At 72 hours : 100 x (Concentration at 48 hours post-randomization-Concentration at randomization)/ Concentration at randomization At 96 hours : 100 x (Concentration at 48 hours post-randomization-Concentration at randomization)/ Concentration at randomization
Area under the concentration curve up to the 96 th hour expressed as a percentage of the concentration at randomization | 96 hours post-randomization
  All concentrations up to the 96th hour post-randomization will be used to generate the area under the curve, and this will be reported as percentage of the concentration at randomization
Number of days alive without mechanical ventilation for 28 days post-randomization | 28 days post randomization
  Patients who leave the hospital after extubation and before the 28th day of randomization will be considered as being free of mechanical ventilation from extubation to the 28th day post randomization
Number of days alive out of critical care for 28 days post-randomization | 28 days post randomization
  This will be defined as the interval from the moment the patient is ready to leave the intensive care until the 28th day of randomization. This will avoid lengthening the theoretical duration of ICU stay due to lack of ward beds
The number of vomiting episodes | through the study complétion, an average of 7 days
  The polyethylene glycol and activated charcoal may induce vomiting, therefore the number of vomiting episodes will be recorded and compared between groups
Number of ventilator-associated pneumonias | through the study complétion, an average of 7 days
  Number of pneumonias occurring through the study completion, an average of 7 days
Number of episodes of upper abdominal pain | through the study complétion, an average of 7 days
  Polyethyleneglycol may cause upper abdominal pain, therefore the number of upper abdominal pain episodes will be recorded and compared between groups
Number of episodes of diarrhoea | through the study complétion, an average of 7 days
  Diarrhea is a therapeutic effect of the polyethylene glycol, therefore the number of diarrhea episodes will be recorded and compared between groups
Presence of hypersensitivity reactions | through the study complétion, an average of 7 days
  Polyethylene glycol may cause allergic reactions such as anaphylactic shock, angioedema, urticaria, rash and pruritus, therefore the presence of allergic reactions will be recorded and compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Voicu Sebastian, MD, Principal Investigator — APHP(ASSISTANCE PUBLIQUE DES HOPITAUX DE PARIS)
Locations (1):
- Sebastian Voicu, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided